CLINICAL TRIAL: NCT01312012
Title: The Effectiveness and Feasibility of Using Antiviral Therapy in Pregnant Women to Reduce Mother-to-infant Transmission of Hepatitis B Virus-drug Test and Follow-up Study
Brief Title: The Antiviral Therapy in Pregnant Women to Reduce Mother-to-infant Transmission of Hepatitis B Virus-drug Test
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201010078M, 201507025RINC
Record Dates: First submitted 2011-01-20; First posted 2011-03-10 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis B Virus Infection, Pregnancy
Keywords: hepatitis B virus,mother-infant transmission, nucleoside analog,pregnant women
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The effectiveness and feasibility, using antiviral therapy (Experimental): Experimental: Subjects receive tenofovir disoproxil fumarate (TDF) oral use prior to delivery in pregnant women with positive serum HBeAg and HBsAg and high HBV DNA levels > 10^8copies / mL, to reduce the rate of mother to infant transmission of HBV infection, and also to monitor the safety of the therapy.
  Interventions: Drug: antiviral therapy
- Control (No Intervention): Subjects receive no intervention, but with blood tests for mothers and infants before and after delivery, as a comparative group to experimental arm.

INTERVENTIONS:
Drug: antiviral therapy — 100-120 pregnant women seropositive for both HBeAg and HBsAg and with hepatitis B viral DNA level > 10 8 copies/mL. Among them, 55-65 pregnant women will receive TDF therapy 300 mg once daily, starting from the gestational age 30-32 (the 3rd trimester) until 4 weeks after delivery of the neonate under informed consent. The total treatment duration will be 3-4 months. Another 45-55 pregnant women with the same serum HBAg and HBsAg and HBV DNA status will be enrolled as the control group with no TDF therapy ( An open-labeled study)
  Arms: The effectiveness and feasibility, using antiviral therapy

SUMMARY:
Since the implementation of universal vaccination in 1984, the chronic HBV carier rate in our general population reduced from 15-20%, down to < 1% in the post-vaccination population. However, children born to HBeAg positive mothers still may be infected with HBV despite immunization. To further reducing the HBV infection in our people, strategies in reducing infection rate in this high risk group are mandatory. Previous small scale studies using lamivudine treatment in pregnant woman in the third trimester has proved effective in reducing children infection rate. The aims of the present study are to conduct a clinical trial in using Tenofovir (category B) to reduce mother-to-infant transmission, and to monitor the hepaitits B viral status and mother hepatitis occurrence. The clinical trials will screen cases of HBsAg positive pregnant women aged 20 to 40 years at gestational at 20-32 weeks. They will be tested for HBsAg and HBeAg. In whom both markers are positive, HBV viral load will be tested. An estimated 180 pregnant women with high HBV viral load (>10^8 copies/mL) will be recruited in the study; including 80-100 subjects treated with Tenofovir 300 mg daily starting from 30-32 weeks of gestation (3rd trimester) and continued to 1 month after delivery; and 80-100 pregnant women are enrolled as controls with no drug given to the mother. The newborn babies are given with HBIG within 24 hours after delivery, and HBV vaccines at 0, 1 and 6 months. Maternal complete blood count (CBC) data tested in the first prenatal examination will be recorded. Plasma AST、ALT levels and HBV DNA are tested before Tenofovir treatment, 1 month after treatment, at the time of delivery, and at 1, 2, 4 and 6 months after delivery. HBsAg、HBeAg、anti-HBs and AST、ALT are tested in the children at day 1, 6 moths and 1 year after birth. The primary outcome is reduction of the HBsAg carrier rate of the children at 6 months of age. The secondary outcome is HBsAg carrier rate of the children at 12 months of age, the change of liver function, HBeAg, and viral load in pregnant mother after treatment.

A follow-up study for investigating safety of mothers and children that has been exposed to maternal tenofovir disoproxil fumarate (TDF) during pregnancy in reducing mother-to-infant hepatitis B virus (HBV) transmissions is conducted. The follow-up study included mother-children pairs 2-4 years after delivery of the children.

ELIGIBILITY:
Inclusion Criteria:

- pregnant women in 30 to 32 weeks of gestation, with positive HBsAg and HBeAg,serum viral load above 8log10 copies per mL

Exclusion Criteria:

* major systemic disease
* Pregnant woman with infection of human immunodeficiency virus or hepatitis C virus
* Pregnant woman is receiving any drug with antiviral activity or any form of drug therapy for hepatitis B virus
* Pregnant woman whose ultrasonographic examination reveals congenital anomaly of the fetus
* Pregnant woman whose amniocentesis reveals any genetic abnormality

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Child-HBsAg | 6 months after delivery
  serum status of HBsAg of the infants at 6 months old( >180 days).

SECONDARY OUTCOMES:
Child HBsAg | 12 months after birth
  Serum HBsAg positivity of the infants at 12 months old, to see whether this child indeed becomes a chronic carrier of HBV.
Children growth parameters | 0-5 years after birth
  body weight and length Z score according to age
Children HBV status | 0-5 years after birth
  HBsAg and anti-HBs positivity rates
Children serum biochemistry | 0-5 years after birth
  Rates of abnormal levels of serum ALT(U/L), creatinine (mg/dL) and calcium (mmol/L)
Maternal HBeAg seroconversion rate | delivery to 5 years after delivery
  Maternal HBeAg seroconversion rate, the time of HBeAg (+) to convert to HBeAg(-) after delivery
Maternal ALT elevation | delivery to 5 years after delivery
  The extent (folds of upper limit of normal, ULN) of ALT elevation and duration.
Maternal HBV DNA | delivery to 5 years after delivery
  Change of levels of HBV DNA (log IU/mL) from baseline
Children bone growth | 2-5 years after birth
  comparisons of BAP levels(U/L) and bone density (DEXA) between control and treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwei Chang, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu HY, Chen HL, Chiang CL, Lai MW, Mu SC, Wen WH, Cheng SW, Hu JJ, Chang KC, Lee CN, Liu CJ, Wu JF, Ni YH, Chang MH; Taiwan Study Group for the Prevention of Mother-to-Infant Transmission of HBV (PreMIT study). Characterization of Hepatitis B Virus in Tenofovir-Treated and Untreated Chronically Infected Mothers and Their Immunoprophylaxis Failure Infants. Clin Infect Dis. 2023 Feb 8;76(3):e783-e790. doi: 10.1093/cid/ciac539. PMID 35789261
- [Derived] Wen WH, Chen HL, Shih TT, Wu JF, Ni YH, Lee CN, Zhao LL, Lai MW, Mu SC, Tung YC, Hsu HY, Chang MH; Taiwan Study Group for the Prevention of Mother-to-Infant Transmission of HBV (PreMIT study)(double dagger). Long-term growth and bone development in children of HBV-infected mothers with and without fetal exposure to tenofovir disoproxil fumarate. J Hepatol. 2020 Jun;72(6):1082-1087. doi: 10.1016/j.jhep.2020.01.021. Epub 2020 Feb 8. PMID 32044401
- [Derived] Chang KC, Chang MH, Lee CN, Chang CH, Wu JF, Ni YH, Wen WH, Shyu MK, Lai MW, Chen SM, Hu JJ, Lin HH, Hsu JJ, Mu SC, Lin YC, Liu CJ, Chen DS, Lin LH, Chen HL; Taiwan Study Group for the Prevention of Mother-to-Infant Transmission of HBV (PreMIT study). Decreased neonatal hepatitis B virus (HBV) viremia by maternal tenofovir treatment predicts reduced chronic HBV infection in children born to highly viremic mothers. Aliment Pharmacol Ther. 2019 Aug;50(3):306-316. doi: 10.1111/apt.15321. Epub 2019 Jul 4. PMID 31271463